CLINICAL TRIAL: NCT06817135
Title: Effect of Scapular Stabilization Exercise on Breastfeeding Women with Non-specific Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saadyya Ahmed Abdalhamed Aladawi (Other)
Responsible Party: Sponsor-Investigator, Saadyya Ahmed Abdalhamed Aladawi, ِِِAssistant Lecturer in the of Women's Health Department, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: scapular stabilization ex.
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Neck Pain
Keywords: scapular stabilization exercise; Breast feeding women
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: The control group got the standard physical therapy program, muscle energy technique for the sternocleidomastoid, elevator scapulae, upper trapezius, and pectoralis major, and advice, while the experimental group got the same conventional physical therapy program in addition to scapular stabilization exercises.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): Got a standard physical therapy program, muscle energy technique for (sternocleidomastoid, elevator scapulae, upper trapezius and pectoralis major) and advice
  Interventions: Other: Muscle Energy Technique; Other: Advice about the right the breastfeeding ergonomic.
- Experimental group (Experimental): got the same conventional physical therapy program plus scapular stabilization exercises.
  Interventions: Other: scapular stabilization exercises; Other: Muscle Energy Technique; Other: Advice about the right the breastfeeding ergonomic.

INTERVENTIONS:
Other: scapular stabilization exercises — Cools exercise using the Thera-Band, including sidelying external rotation, side-lying forward flexion, prone horizontal abduction with external rotation, and prone extension exercises to promote lower trapezius and middle trapezius activity with minimal activation of the upper trapezius part.
  Arms: Experimental group
Other: Muscle Energy Technique — Muscle Energy Technique for the 1.sternocleidomastoid 2. levator scapulae 3. upper trapezius 4. pectoralis major Through mild isometric contractions, it uses the intrinsic energy of a muscle to lengthen it and induce relaxation through autogenic inhibition.
  Other Names: Autogenic Inhibition; Post Isometric Relaxation
Other: Advice about the right the breastfeeding ergonomic. — The patients sit with their backs supported with pillows. Don't lean over the infant. Keep the arms supported and feet on the ground.

SUMMARY:
The purpose of this study is to determine whether scapular stabilization exercises can help breastfeeding women with non-specific neck pain by reducing their neck pain, cervical range of motion, and neck disability index.

DETAILED DESCRIPTION:
The best infant feeding practice is breastfeeding, which has both immediate and long-term advantages for mothers, babies, the environment, the economy, and society as a whole. Mothers who are nursing frequently experience neck pain. Because the scapula and neck are closely related, scapular stabilization is becoming more and more popular for patients with neck pain.

ELIGIBILITY:
Inclusion Criteria:

1. exclusive breastfeeding mothers with immediate to 6-month-old infants.
2. The bilateral cradle position is employed by patients when nursing.
3. Patients had mechanical neck pain.
4. Patients with a body mass index below 30 kg/m²
5. Patients have moderate pain intensity, ranging from 3 to 7 on the visual analogue scale
6. The patients' scores on the Neck Disability Index ranged from 10 to 40 out of 50.

Exclusion criteria:

1. Patients had preterm babies or low-birth-weight babies.
2. pregnant patients
3. Patients had postpartum complications.
4. Patients had inflammation, infection, severe degeneration, congenital deformity, and trauma.
5. Patients had sensory abnormalities or a positive motor reflex.
6. Patients had cancer, metabolic, or systemic diseases.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — breastfeeding mothers
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
functional neck disability | at beginning of the study and after four weeks of treatment
  The Arabic version of the Neck Disability Index Questionnaire (NDI) is used to assess the functional neck disability. It consists of 10 items; each item scores from 0 to 5, where a score of 0 indicates no limitation and a score of 5 indicates maximum limitation.
neck pain intensity | at beginning of the study and after four weeks of treatment
  The Visual Analog Scale VAS was used to assess neck pain intensity for both groups at the beginning of the study and after four weeks of treatment. It is a 10 cm line. 0 means no paint and 10 means maximum pain and the patient chooses a point on the line which reflects the pain

SECONDARY OUTCOMES:
pressure pain threshold | at beginning of the study and after four weeks of treatment
  The local pressure pain threshold over the upper trapezius was measured using a pressure algometer. It is a portable digital algometer that responds linearly to force applications between 0 and 1300 kPa, or roughly 0 and 14 kg. With a 1-cm² circular rubber tip, the device measures the maximum force applied before the subject verbally indicates that the pain threshold has been reached.
cervical range of motion | at beginning of the study and after four weeks of treatment
  The cervical range of motion (flexion, extension, lateral flexion (Rt & Lt), and rotation (Rt & Lt)) is measured with a universal goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Amel M. Yousef, Prof., Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy/ Cairo University, Giza, Dokki, Egypt

REFERENCES:
- [Background] Abd El-Azeim AS, Mahmoud AG, Mohamed MT, El-Khateeb YS. Impact of adding scapular stabilization to postural correctional exercises on symptomatic forward head posture: a randomized controlled trial. Eur J Phys Rehabil Med. 2022 Oct;58(5):757-766. doi: 10.23736/S1973-9087.22.07361-0. Epub 2022 Jun 8. PMID 35673945
- [Background] Nitayarak H, Charntaraviroj P. Effects of scapular stabilization exercises on posture and muscle imbalances in women with upper crossed syndrome: A randomized controlled trial. J Back Musculoskelet Rehabil. 2021;34(6):1031-1040. doi: 10.3233/BMR-200088. PMID 34151819
- See also: Combined effect of graded Thera-Band and scapular stabilization exercises on shoulder adhesive capsulitis post-mastectomy. — https://doi.org/10.1007/s00520-023-07641-6